CLINICAL TRIAL: NCT02151539
Title: Prospective Outcomes of Second-Line Therapy in Acute Graft-Versus-Host Study Including ECP (POSTAGE)
Acronym: POSTAGE
Status: Terminated | Type: Observational
Why Stopped: Low accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Madan Jagasia, MD, Principal Investigator, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC BMT 1401; NCI-2014-01026 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); VICC BMT 1401 (Other: Vanderbilt-Ingram Cancer Center); P30CA068485 (NIH)
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Observational (medical chart review): Study data are collected and managed using REDCap tools at baseline and on days 5, 28, and 56.
  Interventions: Other: medical chart review; Other: quality-of-life assessment

INTERVENTIONS:
Other: medical chart review — Ancillary studies
  Other Names: chart review
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This research trial studies medical chart review in determining outcomes of second-line therapy in patients with acute graft-versus-host disease previously treated with extracorporeal photopheresis or other systemic therapies. Gathering information about second-line therapy in patients with acute graft-versus-host disease may help doctors learn more about the disease and find better treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine 6-month freedom from treatment failure for second-line therapy for acute graft versus host disease (aGVHD).

II. To show that extracorporeal photopheresis (ECP) is associated with a superior 6 month (m) freedom from treatment failure (FFTF) as compared to other treatment modalities for second line therapy for aGVHD.

III. To describe health care burden in patients receiving second line therapy for acute GVHD.

IV. Quality of life measurement using Functional Assessment of Cancer Therapy-Bone Marrow Transplant (FACT-BMT) in patients receiving second line therapy for aGVHD.

OUTLINE:

Study data are collected and managed using Research Electronic Data Capture (REDCap) tools at baseline and on days 5, 28, and 56.

After completion of study, patients are followed up at 6 months, and 1 and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment on study is within 5 days (including weekends) of starting second-line therapy
* aGVHD grade 2 or higher at time of enrollment; patients with late acute and recurrent aGVHD are permitted
* Donor lymphocyte induced aGVHD is permitted ONLY IF donor lymphocyte infusion given for mixed chimerism and not for progression of disease and meeting all other inclusion and exclusion criteria will be eligible
* Corticosteroid refractory or corticosteroid dependent aGVHD

  * Corticosteroid refractory aGVHD is defined as worsening of aGVHD after 3 days of systemic corticosteroids (minimum dose of 1 mg/kg), or no improvement after 7 days of systemic corticosteroids (minimum dose of 1 mg/kg)
  * Corticosteroid dependent aGVHD is defined as recurrence of aGVHD (grade 2 or higher) during corticosteroid taper and prior to reaching 50% of initial starting dose of corticosteroids
* Informed consent form

Exclusion Criteria:

* Has received corticosteroids at 2 mg/kg or higher for 3 weeks or longer as part of first-line therapy for aGVHD
* Has received systemic therapy other than corticosteroids for treatment of aGVHD as part of first-line therapy for acute GVHD; simultaneous uses of topical or enteric corticosteroids or psoralen plus ultraviolet A (PUVA) for first-line are permitted
* aGVHD after second hematopoietic cell transplantation (HCT) is excluded
* Karnofsky performance status =< 50%
* Requiring mechanical ventilation or renal replacement therapy at the time of enrollment
* Histologic or flow-cytometric evidence of relapse or progression of underlying disease; molecular or cytogenetic presence of disease is permitted; mixed chimerism is permitted
* Current or prior diagnosis of chronic GVHD (classic or overlap) as defined by National Institutes of Health (NIH) consensus criteria
* Donor lymphocyte infusion (DLI)-induced aGVHD when DLI was given for progression of the underlying disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study targets patients with acute graft-versus-host disease previously treated with extracorporeal photopheresis or other systemic therapies. Patients can be enrolled by all participating locations.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2014-08-29 (Actual); Primary Completion 2018-10-11 (Actual); Study Completion 2018-10-11 (Actual)

PRIMARY OUTCOMES:
6-month freedom from treatment failure, defined as a patient being alive, without relapse of underlying disease, and without the addition of new systemic therapy for the treatment of aGVHD, within 6 months of starting second line therapy | 6 months
  Rates of 6 m FFTF will be estimated by subtracting rates of total failures from 100%.
Cumulative incidence estimates of relapse | Up to 2 years
  Cox regression models will be used to identify risk factors for failure.
Cumulative incidence estimates of non-relapse mortality | Up to 2 years
  Cox regression models will be used to identify risk factors for failure.
Treatment change as causes of failure during second line treatment | Up to 2 years
  Cox regression models will be used to identify risk factors for failure.
Health care burden in patients receiving second line therapy for acute GVHD | Up to 6 months
  The incremental budget spend between the patients receiving treatment with ECP and patients receiving other modalities will be measured and economic methods will be used to calculate an incremental cost effectiveness ratio for relevant clinical end points. Health economic data relating to hospitalizations (length of stay in myelosuppressive unit, high-dependency unit [step-down unit], intensive care unit), high cost drugs, total parenteral nutrition and surgical procedures will also be collected allowing comparisons to be made between patients treated with ECP and other treatment options.
Quality of life measured using FACT-BMT | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Madan Jagasia, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (7):
- United States (4):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic, Rochester, Minnesota
  - The Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt-Ingram Cancer Center (VICC), Nashville, Tennessee
- Medical University Vienna, Vienna, Austria
- Klinikum der Universität Regensburg, Regensburg, Germany
- Nottingham City Hospital, Nottingham, United Kingdom

REFERENCES:
- See also: Vanderbilt-Ingram Cancer Center, Find a Clinical Trial — http://www.vicc.org/ct/